CLINICAL TRIAL: NCT02473822
Title: ACL Reconstruction With the TLS Technique (Tape Locking Screw) and Return to Sport: Serial 5-year Independent Designers
Brief Title: ACL Reconstruction With the TLS Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-24
Record Dates: First submitted 2015-05-14; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Joint Trauma
Keywords: anterior cruciate ligament; Tape Locking Screw; LCA; joint trauma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-interventional study to retrospectively validate the technical use TLS (Tape Locking Screw) in the anterior cruciate ligament. The investigators goal is to test the validity of the technique and its positive influence on the resumption of sporting activities in relation to the existing literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients operated in the service in 2014 to care for end-stage knee osteoarthritis by implantation of a total knee prosthesis.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing care of knee instability in chronic laxity of anterior cruciate ligament by ligament according to TLS technique.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Resumption of sporting activities | every 3 months over a period of one year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France